CLINICAL TRIAL: NCT00776204
Title: The Optical Coherence Tomography Drug Eluting Stent Investigation(OCTDESI)
Brief Title: The Optical Coherence Tomography Drug Eluting Stent Investigation
Acronym: OCTDESI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Labcoat, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBCT-H03-07
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug eluting stent; Percutaneous Coronary Interventions; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Drug Eluting Stent
  Interventions: Device: JACTAX Drug eluting stent
- 2 (Active Comparator): Drug Eluting Stent
  Interventions: Device: JACTAX LD drug eluting stent
- 3 (Active Comparator): Drug Eluting Stent
  Interventions: Device: Taxus Libertè

INTERVENTIONS:
Device: JACTAX Drug eluting stent — Jactax stent placed in coronary artery
  Other Names: JACTAX Drug eluting stent (Labcoat Ltd, Galway, Ireland)
  Arms: 1
Device: JACTAX LD drug eluting stent — JACTAX LD stent placed in coronary artery
  Other Names: JACTAX LD Drug eluting stent (Labcoat Ltd, Galway, Ireland)
  Arms: 2
Device: Taxus Libertè — Taxus Libertè stent placed in coronary artery
  Other Names: Taxus Libertè (Boston Scientific, Natick, MA)
  Arms: 3

SUMMARY:
The objective of this study is to evaluate the completeness of struts coverage and vessel wall response to the new generation JACTAX drug-eluting stent vs Taxus stent in de novo coronary artery lesions at 6 months post index procedure. To investigate the completeness of the coverage as well as the number of uncovered stent struts per section, high resolution (~ 10-15 µm axial) intracoronary Optical Coherence Tomography (OCT) will be used.

DETAILED DESCRIPTION:
The risk of late stent thrombosis represents a major concern for patients treated with first generation drug-eluting stents (DES). Delayed healing and poor endothelialization are common findings in vessels treated with DES and are probably related to the amount of drug and polymer applied to a DES. There is evidence to suggest that polymer applications may influence the processes of inflammation and vessel healing. The JACTAX family of DES have been designed to provide a maximum amount of drug delivered directly to coronary vessel tissue while excluding polymer and drug from contact within the vessel lumen. The JACTAX stents are comprised of a currently marketed bare metal stent (Libertè™) coated exclusively on the ablumenal stent surface with a carrier containing a bioerodable polymer, Polylactide and paclitaxel. The objective of this prospective study is to measure the completeness of strut coverage and vessel wall response (strut malapposition, neointima disomogeneities in texture) to the JACTAX stents vs Taxus Libertè in de novo coronary artery lesions at 6 months post index procedure. Optical Coherence Tomography (OCT) that detects smaller degrees of stent strut coverage more accurately than IVUS will be used at 6 months follow-up. Intravascular ultrasound (IVUS) will be performed as per normal practice at any index procedures and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Patient is ≥ 18 years of age
2. Patient is eligible for percutaneous coronary intervention (PCI)
3. Patient demonstrates a left ventricular ejection fraction (LVEF) of ≥ 25%
4. Patient or legal guardian understands and agrees to comply with all specified study requirements and provides written Informed Consent to this effect.

Angiographic Inclusion Criteria

1. Target lesion is de novo native coronary artery lesion (i.e., a coronary lesion not previously treated) ≤ 25 mm that can be treated with a single JACTAX, JACTAX LD or TAXUS stent
2. A second lesion in a second vessel may be treated with one (1) TAXUS™ Libertè™ DES or a bare metal stent.

Exclusion Criteria:

General Exclusion Criteria

1. The patient has a life expectancy of less than 24 months due to another medical condition
2. Patient has a history of hypersensitivity to paclitaxel or structurally related compounds
3. Patient exhibits cardiogenic shock (systolic pressure < 80mm Hg and PCWP > 20mm Hg or cardiac index <1.8 liters/minute/m2 or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure>80 mm Hg) for any time within 24 hours prior to index procedure
4. Patient demonstrates evidence of acute or chronic renal dysfunction (serum creatinine > 2.0 mg/dl or177 µmol/l)
5. Planned cardiac surgery procedure ≤ 6 months post-index procedure
6. Patient demonstrates evidence of a acute myocardial infarction (eg. STEMI or enzyme elevation CK > 2X local laboratory's ULN unless CK-MB is < 2X ULN) 7) Cerebrovascular accident (CVA) including stroke or TIA within previous 3 months
7. Patient demonstrates evidence of leukopenia (leukocyte count < 3.5 X 109/liter)
8. Patient demonstrates evidence of thrombocytopenia (platelet count < 100,000/mm3) or thrombocytosis (>750,000/mm3)
9. Patient is contraindicated to ASA (successful prior desensitization to ASA is not an exclusion), clopidogrel, or ticlopidine
10. Patient is currently on warfarin, or possibility of treatment with warfarin during the following 6 months post index procedure
11. Patient has been treated with paclitaxel or other chemotherapeutic agents within 12-months prior to planned index procedure
12. Anticipated treatment with paclitaxel or oral rapamycin during any period in the 6-months after the index procedure
13. Patient has received a drug eluting stent within 12-months prior to planned index procedure
14. Previous or planned treatment with intravascular brachytherapy in target vessel
15. Known allergy to stainless steel
16. Female or male with known intention to procreate within 3 months after the index procedure (due to the exposure to paclitaxel and unknown affect it may have on the fetus)
17. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the 9 months post index procedure
18. Patient that in the opinion of the investigator is not clinically appropriate for OCT evaluation.

Angiographic Exclusion Criteria

1. Evidence of thrombus of the study vessel, based on angiography or IVUS
2. Study lesion is totally occluded (TIMI flow ≤ 1) either at baseline or before pre-dilatation
3. Study lesion, or the study vessel proximal to the study lesion is moderately or severely calcified, by visual estimate
4. Study lesion is ostial in location (within 3.0 mm of vessel origin)
5. Study lesion involving arterial segments with highly tortuous anatomy or where lesion is located within or distal to a >60 degree bend in the vessel
6. Study lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel > 2.0 mm in diameter
7. Left main coronary artery disease (stenosis >50%) whether protected or unprotected
8. Target lesion length > 25 mm, based on visual estimate by operator
9. Target vessel diameter > 3.5 mm, based on visual estimate by operator
10. Target vessel diameter < 2.75 mm based on visual estimate by operator
11. Pre-treatment of the target lesion (excluding predilation) with another interventional device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of stent struts uncovered and/or malapposed at OCT | 6 months

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 12 and 24 months
Stent Thrombosis | 12 and 24 months
Target Lesion Revascularization | 12 and 24 months
Procedural success | through discharge
QCA parameters: mean lumen diameter, acute gain, late loss and binary restenosis (≥ 50% diameter stenosis) rate | 6 months
IVUS parameters: neointimal area volume, stent and area volumes, stent apposition, and percent net volume obstruction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Ospedali Riuniti di Bergamo, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luscher TF, Steffel J, Eberli FR, Joner M, Nakazawa G, Tanner FC, Virmani R. Drug-eluting stent and coronary thrombosis: biological mechanisms and clinical implications. Circulation. 2007 Feb 27;115(8):1051-8. doi: 10.1161/CIRCULATIONAHA.106.675934. PMID 17325255
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Kang WC, Han SH, Choi KR, Ahn TH, Shin EK. Acute myocardial infarction caused by late stent thrombosis after deployment of a paclitaxel-eluting stent. J Invasive Cardiol. 2005 Jul;17(7):378-80. No abstract available. PMID 16003026
- [Background] Virmani R, Liistro F, Stankovic G, Di Mario C, Montorfano M, Farb A, Kolodgie FD, Colombo A. Mechanism of late in-stent restenosis after implantation of a paclitaxel derivate-eluting polymer stent system in humans. Circulation. 2002 Nov 19;106(21):2649-51. doi: 10.1161/01.cir.0000041632.02514.14. PMID 12438288
- [Background] Carter AJ, Aggarwal M, Kopia GA, Tio F, Tsao PS, Kolata R, Yeung AC, Llanos G, Dooley J, Falotico R. Long-term effects of polymer-based, slow-release, sirolimus-eluting stents in a porcine coronary model. Cardiovasc Res. 2004 Sep 1;63(4):617-24. doi: 10.1016/j.cardiores.2004.04.029. PMID 15306217
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Background] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Background] Guagliumi G, Sirbu V. Optical coherence tomography: high resolution intravascular imaging to evaluate vascular healing after coronary stenting. Catheter Cardiovasc Interv. 2008 Aug 1;72(2):237-47. doi: 10.1002/ccd.21606. PMID 18655155
- [Derived] Guagliumi G, Sirbu V, Musumeci G, Bezerra HG, Aprile A, Kyono H, Fiocca L, Matiashvili A, Lortkipanidze N, Vassileva A, Popma JJ, Allocco DJ, Dawkins KD, Valsecchi O, Costa MA. Strut coverage and vessel wall response to a new-generation paclitaxel-eluting stent with an ultrathin biodegradable abluminal polymer: Optical Coherence Tomography Drug-Eluting Stent Investigation (OCTDESI). Circ Cardiovasc Interv. 2010 Aug;3(4):367-75. doi: 10.1161/CIRCINTERVENTIONS.110.950154. Epub 2010 Jul 20. PMID 20647562